CLINICAL TRIAL: NCT01971021
Title: Vascular Access in Cancer Patients - PICC vs PORT in a Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Ryhov County Hospital (Other)
Responsible Party: Principal Investigator, Knut Taxbro, MD Consultant in Anesthesia and Intensive Care, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EPN Linkoping 2013/56-31
Record Dates: First submitted 2013-09-24; First posted 2013-10-28 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Focus of Study
MeSH Terms: interventions — Catheterization, Peripheral

STUDY DESIGN:
Intervention Model Description: open label pragmatic
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PICC-line (Active Comparator): PICC line insertion.
  Interventions: Device: PICC or subcutaneous venous port
- PORT (Active Comparator): Subcutaneous venous port insertion
  Interventions: Device: PICC or subcutaneous venous port

INTERVENTIONS:
Device: PICC or subcutaneous venous port

SUMMARY:
As of today there is very limited scientific knowledge in whicj of the two vascular access devices (PICC-line or venous ports) that offers the lowest complicationrates in cancerpatients. The study group wants to clearify this unsolved matter by comparing the two systems. Our primary endpoint is the presens of catheter related venous thrombosis. We are also looking at all catheter related complications and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* cancer treatment with need for central venous access
* Age >18 yrs
* Suspected survival > 4 weeks
* Need of central venous access >4 weeks

Exclusion Criteria:

* Ongoing uncontrolled systemic infection
* Prescence of significant thrombosis/stenosis in arm or central veins
* Unability to communicate
* Probable upcoming need for dialysis fistula

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
The occurence of catheter related venous thrombosis | Upon clinical suspiscion during the one the patient i enrolled in the study
  regular follow-ups at month 1, 3, 6 and 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Oncology, Jönköping, Sweden

REFERENCES:
- [Derived] Utas A, Seifert S, Taxbro K. Peripherally inserted central catheters versus implanted port catheters in patients with breast cancer: a post hoc analysis of the PICCPORT randomised controlled trial. BJA Open. 2025 Feb 4;13:100377. doi: 10.1016/j.bjao.2025.100377. eCollection 2025 Mar. PMID 39991709
- [Derived] Taxbro K, Hammarskjold F, Juhlin D, Hagman H, Bernfort L, Berg S. Cost analysis comparison between peripherally inserted central catheters and implanted chest ports in patients with cancer-A health economic evaluation of the PICCPORT trial. Acta Anaesthesiol Scand. 2020 Mar;64(3):385-393. doi: 10.1111/aas.13505. Epub 2019 Nov 27. PMID 31721153
- [Derived] Taxbro K, Hammarskjold F, Thelin B, Lewin F, Hagman H, Hanberger H, Berg S. Clinical impact of peripherally inserted central catheters vs implanted port catheters in patients with cancer: an open-label, randomised, two-centre trial. Br J Anaesth. 2019 Jun;122(6):734-741. doi: 10.1016/j.bja.2019.01.038. Epub 2019 Apr 17. PMID 31005243